CLINICAL TRIAL: NCT01449500
Title: Effect of Dietary Supplementation With L. Reuteri ProGastria in H. Pylori-infected Adult Subjects Treated Only With Proton Pump Inhibitors
Brief Title: Supplementation With L. Reuteri in H. Pylori Infected Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lama Medical Care s.r.o. (Industry)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CSUB0028
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Dyspepsia; H. Pylori Infection
Keywords: Dyspeptic H.pylori-infection
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- L. reuteri (Active Comparator): L. reuteri will be delivered at a dose of 1x108 CFU of each strain of L. reuteri giving a final dose of L. reuteri of 2x108 CFU. One dose is to be taken once per day giving a dose of L. reuteri of 2x108 CFU/day.
  Intervention: Dietary Supplement: L. reuteri DSM 17938 and ATCC PTA 6475
  Interventions: Dietary Supplement: L. reuteri

INTERVENTIONS:
Dietary Supplement: L. reuteri — Chewable tablet, one tablet/day for 28 days
  Other Names: L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475
  Arms: L. reuteri
Dietary Supplement: Placebo — Chewable tablet, one tablet per day for 28 days
  Arms: Placebo

SUMMARY:
To determine whether simultaneous use of L. reuteri ProGastria and proton pump inhibitors can eradicate H. pylori in humans in the absence of antibiotics.

DETAILED DESCRIPTION:
Fifty-six (56) subjects, aged 18-70 years will be recruited from patients with dyspeptic symptoms referred to the clinic for consultation about H. pylori infection and who have not previously been treated for this infection. Patients in whom H. pylori infection is confirmed (by endoscopy with biopsy) and who fulfil the inclusion criteria, will be invited to enter the study. After written consent has been obtained subjects will be randomly allocated to one of two groups, one to receive omeprazole (2x20mg/day) + 1 tablet placebo per day and the other to receive omeprazole (2x20mg/day) + 1 tablet (2x108 CFU L. reuteri) ProGastria per day.

After randomisation on Day 0 of the study, the subjects will also be asked to complete a gastrointestinal symptom rating score (GSRS) to determine baseline symptomology.

Intervention will begin on Day 1 and last for 28 days after which therapy will be stopped. The subjects will be asked to complete the GSRS questionnaire on Day 14 and Day 28. At Day 14, the patients GSRS scores are monitored and the patients interviewed. In those patients where there is a marked deterioration of their condition or symptoms, these will be considered treatment failures and eradication therapy will then be started on Day 15.

The day after therapy is stopped (Day 29), patients symptoms will be assessed. All patients will undergo gastroscopy to determine the presence of H. pylori or not. If H. pylori infection is confirmed (by endoscopy and biopsy staining), these subjects will be given triple therapy to eradicate the infection and followed up on Day 90 of the study.

On Day 29, those patients that no longer complain of symptoms and are shown to be free of H. pylori infection by endoscopy (treatment success group), will continue with no further therapy until Day 90.

On Day 90 all subjects will be given a UBT to determine the presence of H. pylori infection and symptoms will be again assessed using GSRS. Asymptomatic patients with negative breath test will be considered recovered. In those patients where persistent H. pylori infection is confirmed by breath test, second line therapy will be implemented as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-70 years
* Infection with H. pylori defined by endoscopic examination with biopsy H. pylori staining
* Non-ulcer dyspepsia
* Absence of other pathology as shown by basic clinical laboratory tests (blood and urine) as well as abdominal ultrasound
* No earlier eradication therapy for H. pylori infection
* Written informed consent
* Stated availability throughout the entire study period
* Mental ability to understand and willingness to fulfil all the details of the protocol.

Exclusion Criteria:

* Duodenal or gastric ulcer
* MALT lymphoma
* Gastric resection (at any time)
* First level relatives of gastric cancer patients
* Absence of GI symptoms
* Use of NSAIDs, aspirin or other anti-inflammatory drugs within 1 week (for occasional use) or 3 weeks (for chronic use) of inclusion
* Use of oral antibiotics and/or PPIs and/or H2-antagonists during the 2 weeks prior to ingestion of the study product
* Pregnancy
* Participation in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Increase in the number of subjects with treatment success after 28 days of treatment with omeprazole + L. reuteri compared to those given omeprazole + placebo. | 28 days
  Treatment success is defined as the absence of H. pylori infection as shown by a significant reduction in symptoms on Day 28 and by the absence of H. pylori on gastric biopsy at Day 28.

SECONDARY OUTCOMES:
Fewer patients in the L. reuteri treatment success group with demonstrated presence of H. pylori infection, measured as UBT on Day 90 compared to the placebo treatment success group | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ladislav Kuzela, MD, Principal Investigator — Gastroenterology Hepatology Centrum THALION, Poliklinika Mytna - 2.poscodie Mytna ul. 5, 811 07, Bratislava, Slovakia
Locations (1):
- Gastroenterology Hepatology Centrum THALION, Poliklinika Mytna - 2.poscodie Mytna ul. 5, Bratislava, Slovakia